CLINICAL TRIAL: NCT02627924
Title: Real-World Outcome of Rheumatoid Arthritis Patients in Korea on Adalimumab (ROCKA Study)
Brief Title: Real-World Outcome of Rheumatoid Arthritis Patients in Korea on Adalimumab
Acronym: ROCKA
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P15-777
Record Dates: First submitted 2015-12-09; First posted 2015-12-11 (Estimated); Results first posted 2019-03-22 (Actual); Last update posted 2019-03-22 (Actual); Status verified 2018-11

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Work productivity; patient-reported QoL(Quality of Life)
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adalimumab: Participants diagnosed with rheumatoid arthritis who were prescribed adalimumab according to their physician's discretion and routine clinical practice.

SUMMARY:
The study is designed as a prospective, observational study to assess the effect of adalimumab on health-related quality of life (QoL) and work productivity in patients with rheumatoid arthritis (RA) in Korea.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a diagnosis of RA as defined by the 1987 revised American College of Rheumatology (ACR) classification criteria and/or the ACR/the European League against Rheumatism (EULAR) 2010 classification criteria (any duration since diagnosis).
* Male or female subject ≥ 18 years of age (local definition according to adalimumab label) who is in compliance with eligibility for adalimumab based on the local label.
* Patients with moderate to severe RA defined as Disease Activity Score in 28 Joints (DAS28) (ESR) or DAS28 (CRP) > 3.2
* Biologically treatment naïve and initiated adalimumab at baseline visit
* Availability of clinical data of the previous 12 weeks prior to baseline
* Ability to self-complete patient questionnaires
* Subject must be able and willing to provide written informed consent and comply with the requirements of this study protocol.

Exclusion Criteria:

* Patients who are pregnant or breast feeding at enrolment or wish to become pregnant in the next 24 weeks.
* Participation in any RA-related clinical trial at the time of enrolment, at baseline or at any point during the past 24 weeks prior to baseline
* Patients who in the clinician's view, may not be able to accurately report their QoL or prior resource utilization
* Patients who in the clinician's view, may not be able to adhere to adalimumab therapy over 24 weeks.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects receiving Adalimumab with Rheumatoid Arthritis (RA) in Korea
Sampling Method: Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2015-11-18 (Actual); Primary Completion 2017-12-28 (Actual); Study Completion 2017-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — http://rxabbvie.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Ninety-one patients diagnosed with rheumatoid arthritis (RA) were enrolled at nine different sites in Korea.
Period: Overall Study
Arm/Group | Adalimumab
Started | 91
Completed | 79
Not Completed | 12

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 91
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.7 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64
  Male | 27
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Heath Assessment Questionnaire - Disability Index (HAQ-DI) [Mean (Standard Deviation); unit: units on a scale] — The HAQ-DI is a patient-reported assessment of physical function that includes 20 items in eight categories including dressing and grooming, arising, eating, walking, hygiene, reach, grip and common daily activities. Patients were asked about their ability to complete these tasks in the past week using the following categories: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). Scores on each task were summed and averaged to provide an overall score ranging from 0 (best) to 3 (worst), where higher scores represent a high-dependency disability.
  units on a scale | 1.33 (0.73)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Health Assessment Questionnaire - Disability Index (HAQ-DI) Score at Week 24
Description: The HAQ-DI is a patient-reported assessment of physical function that includes 20 items in eight categories representing a comprehensive set of functional activities, including dressing and grooming, arising, eating, walking, hygiene, reach, grip and common daily activities. Patients were asked about their ability to complete these tasks in the past week using the following categories: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). Scores on each task were summed and averaged to provide an overall score ranging from 0 (best) to 3 (worst), with a higher score representing a high-dependency disability.
Time Frame: Baseline and week 24
Population: Participants who were still receiving adalimumab at week 24 and with available HAQ-DI data at baseline and week 24.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 71
units on a scale | -0.67 (0.67)
Statistical Analysis 1: Comparison: Adalimumab; Test type: Other; p < 0.0001, Paired t-test; The mean change was tested with a paired t-test without adjusting for baseline disease severity

2. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire - Disability Index (HAQ-DI) Score at Week 12
Description: as for outcome 1
Time Frame: Baseline and week 12
Population: Participants who were still receiving adalimumab at week 24 and with available HAQ-DI data at baseline and week 12.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 79
units on a scale | -0.46 (0.60)
Statistical Analysis 1: Comparison: Adalimumab; Test type: Other; p < 0.0001, Paired t-test; The mean change was tested with a paired t-test without adjusting for baseline disease severity

3. Secondary Outcome: Percentage of Participants Achieving a Clinically Meaningful Improvement on the HAQ-DI at Weeks 12 and 24
Description: The HAQ-DI is a patient-reported assessment of physical function that includes 20 items in eight categories representing a comprehensive set of functional activities, including dressing and grooming, arising, eating, walking, hygiene, reach, grip and common daily activities. Patients were asked about their ability to complete these tasks in the past week using the following categories: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). Scores on each task were summed and averaged to provide an overall score ranging from 0 (best) to 3 (worst), with a higher score representing a high-dependency disability.
  A clinically meaningful improvement was defined as an improvement of -0.22 points or greater in the HAQ-DI score.
Time Frame: Baseline, week 12 and week 24
Population: Participants still receiving adalimumab and with available data at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 88
percentage of participants
  Week 12: number analyzed (Participants) | 79
  Week 12 | 65.8
  Week 24: number analyzed (Participants) | 71
  Week 24 | 77.5

4. Secondary Outcome: Change From Baseline in Short-Form 36 (SF-36) Physical Component Summary and Mental Component Summary Scores at Weeks 12 and 24
Description: The Medical Outcome Study Short Form 36-Item Health Survey, Version 2 (SF-36) is a self-administered instrument that measures the impact of disease on overall quality of life and consists of 36 questions in eight domains (physical function, pain, general and mental health, vitality, social function, physical and emotional health).
  The summary physical health score included the following subscales: physical functioning, role-physical, bodily pain, and general health. The summary mental health score included the following subscales: vitality, social functioning, role-emotional, and mental health.
  Each score ranges from 0 to 100 where higher scores indicate a better quality of life. A positive change from Baseline score indicates an improvement.
Time Frame: Baseline, week 12, and week 24
Population: Participants still receiving adalimumab and with available data at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 88
units on a scale
  Physical Component Score at Week 12: number analyzed (Participants) | 79
  Physical Component Score at Week 12 | 6.56 (6.98)
  Physical Component Score at Week 24: number analyzed (Participants) | 71
  Physical Component Score at Week 24 | 9.51 (7.77)
  Mental Component Score at Week 12: number analyzed (Participants) | 79
  Mental Component Score at Week 12 | 5.26 (11.62)
  Mental Component Score at Week 24: number analyzed (Participants) | 71
  Mental Component Score at Week 24 | 6.63 (12.31)
Statistical Analysis 1: Comparison: Adalimumab; Change From Baseline in Physical Component Score at Week 12; Test type: Other; p < 0.0001, Paired t-test
Statistical Analysis 2: Comparison: Adalimumab; Change From Baseline in Physical Component Score at Week 24; Test type: Other; p < 0.0001, Paired t-test
Statistical Analysis 3: Comparison: Adalimumab; Change From Baseline in Mental Component Score at Week 12; Test type: Other; p = 0.0001, Paired t-test
Statistical Analysis 4: Comparison: Adalimumab; Change From Baseline in Mental Component Score at Week 24; Test type: Other; p < 0.0001, Paired t-test

5. Secondary Outcome: Change From Baseline in EuroQol 5-Dimension 3-Level (EQ-5D-3L) Index at Weeks 12 and 24
Description: The EQ-5D-5L descriptive system comprises 5 dimensions of health-related quality of life states (mobility, selfcare, usual activities, pain/discomfort, and anxiety/depression) each of which can take one of three responses. The responses record three levels of severity ('no problems', 'some problems', and 'extreme problems') within a particular EQ-5D-3L dimension. The EQ-5D-3L results were converted into a weighted health state index with scores ranging from approximately 0 (death) to 1 (full health). A positive change from baseline indicates improvement.
Time Frame: Baseline, week 12, and week 24
Population: Participants still receiving adalimumab and with available data at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 88
units on a scale
  Week 12: number analyzed (Participants) | 78
  Week 12 | 0.15 (0.24)
  Week 24: number analyzed (Participants) | 70
  Week 24 | 0.18 (0.25)
Statistical Analysis 1: Comparison: Adalimumab; Change from Baseline in EQ-5D-3L at 12 weeks; Test type: Other; p < 0.0001, Paired t-test
Statistical Analysis 2: Comparison: Adalimumab; Change from Baseline in EQ-5D-3L at 24 weeks; Test type: Other; p < 0.0001, Paired t-test

6. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment Questionnaire (WPAI) at Weeks 12 and 24
Description: The Work Productivity and Activity Impairment (WPAI) questionnaire for general health is a validated tool in RA consisting of 6 questions, based on patient recall of the previous 7 days. WPAI assesses work time missed due to illness (absenteeism), impairment at work due to health (presenteeism), overall work impairment due to health (an aggregate measure of both absenteeism and presenteeism), and total non-occupational activity impairment due to health. WPAI scores are expressed as impairment percentages, with higher scores indicating worse outcomes. A negative change from baseline indicates improvement.
Time Frame: Baseline, week 12, and week 24
Population: Participants still receiving adalimumab and with available data at each time point. Overall work impairment was only assessed in participants who were employed.
Measure: Mean (Standard Deviation); unit: percent impairment
Arm/Group | Adalimumab
Number analyzed (Participants) | 88
percent impairment
  Overall Work Impairment at Week 12: number analyzed (Participants) | 24
  Overall Work Impairment at Week 12 | -19 (32)
  Overall Work Impairment at Week 24: number analyzed (Participants) | 20
  Overall Work Impairment at Week 24 | -25 (31)
  Activity Impairment at Week 12: number analyzed (Participants) | 72
  Activity Impairment at Week 12 | -15 (31)
  Activity Impairment at Week 24: number analyzed (Participants) | 65
  Activity Impairment at Week 24 | -25 (34)
Statistical Analysis 1: Comparison: Adalimumab; Change From Baseline in Overall Work Impairment at Week 12; Test type: Other; p = 0.0098, Paired t-test
Statistical Analysis 2: Comparison: Adalimumab; Change From Baseline in Overall Work Impairment at Week 24; Test type: Other; p = 0.0015, Paired t-test
Statistical Analysis 3: Comparison: Adalimumab; Change From Baseline in Activity Impairment at Week 12; Test type: Other; p < 0.0001, Paired t-test
Statistical Analysis 4: Comparison: Adalimumab; Change From Baseline in Activity Impairment at Week 24; Test type: Other; p < 0.0001, Paired t-test

7. Secondary Outcome: Patient Treatment Satisfaction
Description: Participants were asked to answer the following four questions as either Very satisfied, Somewhat satisfied, Neither satisfied nor dissatisfied, Somewhat dissatisfied, or Very dissatisfied.
  Question 1: Satisfaction with RA treatment in improving morning stiffness in and around the joints
  Question 2: Satisfaction with RA treatment improving mobility
  Question 3: Satisfaction with RA treatment improving the ability to perform daily living requiring fine motor skills
  Questions 4: Satisfaction with RA treatment overall
Time Frame: Baseline, week 12 and week 24
Population: Participants still receiving adalimumab and with available data at each time point.
Measure: Count of Participants; unit: Participants
Groups:
- Baseline: Participants who completed the patient treatment satisfaction questionnaire at baseline.
- Week 12: Participants who completed the patient treatment satisfaction questionnaire at week 12
- Week 24: Participants who completed the patient treatment satisfaction questionnaire at week 24.
Arm/Group | Baseline | Week 12 | Week 24
Number analyzed (Participants) | 88 | 79 | 71
Participants
  Question 1 - morning stiffness: Very satisfied | 9 | 27 | 30
  Question 1 - morning stiffness: Somewhat satisfied | 15 | 24 | 19
  Question 1 - morning stiffness: Neither satisfied nor dissatisfied | 26 | 17 | 14
  Question 1 - morning stiffness: Somewhat dissatisfied | 25 | 7 | 6
  Question 1 - morning stiffness: Very dissatisfied | 13 | 4 | 2
  Question 2 - Mobility: Very satisfied | 6 | 27 | 27
  Question 2 - Mobility: Somewhat satisfied | 25 | 24 | 22
  Question 2 - Mobility: Neither satisfied nor dissatisfied | 26 | 18 | 13
  Question 2 - Mobility: Somewhat dissatisfied | 21 | 7 | 7
  Question 2 - Mobility: Very dissatisfied | 10 | 3 | 2
  Question 3 - Fine motor skills: Very satisfied | 12 | 27 | 33
  Question 3 - Fine motor skills: Somewhat satisfied | 12 | 24 | 16
  Question 3 - Fine motor skills: Neither satisfied nor dissatisfied | 25 | 19 | 15
  Question 3 - Fine motor skills: Somewhat dissatisfied | 21 | 7 | 6
  Question 3 - Fine motor skills: Very dissatisfied | 18 | 2 | 1
  Question 4 - Treatment overall: Very satisfied | 9 | 32 | 32
  Question 4 - Treatment overall: Somewhat satisfied | 14 | 22 | 17
  Question 4 - Treatment overall: Neither satisfied nor dissatisfied | 32 | 16 | 16
  Question 4 - Treatment overall: Somewhat dissatisfied | 21 | 7 | 6
  Question 4 - Treatment overall: Very dissatisfied | 12 | 2 | 0

8. Secondary Outcome: Healthcare Resource Utilization: Number of Participants With Visits to Healthcare Professionals for Treatment of Rheumatoid Arthritis
Description: The healthcare resource utilization (HCRU) questionnaire collected data on the healthcare resources used over the course of the study.
Time Frame: 24 weeks
Population: Enrolled participants who did not discontinue adalimumab during the study
Measure: Count of Participants; unit: Participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 88
Participants
  Family medicine | 2
  Rheumatologist | 87
  Orthopaedist | 4
  Internist | 6
  Emergency department | 0
  Traditional Medicine | 3
  Rehabilitation Medicine | 2
  Other | 2
  Any healthcare professional | 87

9. Secondary Outcome: Healthcare Resource Utilization: Number of Participants Who Underwent Procedures Related to Treatment of Rheumatoid Arthritis
Description: as for outcome 8
Time Frame: 24 weeks
Population: Enrolled participants who did not discontinue adalimumab during the study
Measure: Count of Participants; unit: Participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 88
Participants
  Chest X-Ray | 19
  Spine X-Ray | 5
  Neck X-Ray | 2
  Shoulder X-Ray | 4
  Hand X-Ray | 4
  Knee X-Ray | 5
  Magnetic resonance imaging (MRI) | 0
  Computed tomography (CT) scan | 4
  Electrocardiogram | 4
  Blood sample taken | 61
  Urine test | 35
  Endoscopy | 2
  Bone scan | 1
  Liver function test | 8
  Tuberculin Skin Test | 3
  Sputum tests | 2
  Other | 8
  Any Procedure | 67

10. Secondary Outcome: Healthcare Resource Utilization: Number of Participants With Hospitalization Related to Rheumatoid Arthritis
Description: as for outcome 8
Time Frame: 24 weeks
Population: Enrolled participants who did not discontinue adalimumab during the study
Measure: Count of Participants; unit: Participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 88
Participants | 3

11. Secondary Outcome: Healthcare Resource Utilization: Number of Participants With Surgery Related to Rheumatoid Arthritis
Description: as for outcome 8
Time Frame: 24 weeks
Population: Enrolled participants who did not discontinue adalimumab during the study
Measure: Count of Participants; unit: Participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 88
Participants | 0

12. Secondary Outcome: Healthcare Resource Utilization: Number of Participants Who Received Concomitant Medications for Rheumatoid Arthritis
Description: as for outcome 8
Time Frame: 24 weeks
Population: Enrolled participants who did not discontinue adalimumab during the study
Measure: Count of Participants; unit: Participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 88
Participants
  Disease-modifying Antirheumatic Drug (DMARD) | 36
  Anti-inflammatory Drug (NSAID) | 32
  Others | 26
  Any Concomitant Medication | 44

ADVERSE EVENTS:
Time Frame: Up to 34 weeks
Arm/Group | Adalimumab
All-Cause Mortality (participants affected / at risk) | 0/91
Serious Adverse Events (participants affected / at risk) | 6/91
Other Adverse Events (participants affected / at risk) | 6/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab (N=91)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Spinal column stenosis (Nervous system disorders) | 1
Pneumonia bacterial (Infections and infestations) | 1
Deep vein thrombosis (Vascular disorders) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Drug ineffective (General disorders) | 1
Rheumatoid arthritis (Immune system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab (N=91)
Rash (Skin and subcutaneous tissue disorders) | 2
Injection site erythema (General disorders) | 2
Rosacea (Skin and subcutaneous tissue disorders) | 1
Antinuclear antibody increased (Investigations) | 1
C-reactive protein increased (Investigations) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Drug ineffective (General disorders) | 1
Haemoglobin decreased (Investigations) | 1
Injection site pruritus (General disorders) | 2
Injection site rash (General disorders) | 1
Red blood cell sedimentation rate increased (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2017-12-26): https://cdn.clinicaltrials.gov/large-docs/24/NCT02627924/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-02): https://cdn.clinicaltrials.gov/large-docs/24/NCT02627924/SAP_001.pdf